CLINICAL TRIAL: NCT05380934
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial of TQH3821 in Adult Healthy Subjects
Brief Title: A Clinical Trial of Safety and Tolerance of TQH3821 Tablets in Adult Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH3821-I-01
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- TQH3821 Tablets (Single Administration Dose) (Experimental): TQH3821 tablets, Single administration
  Interventions: Drug: TQH3821 tablets
- TQH3821 Placebo Tablets (Single Administration Dose) (Placebo Comparator): TQH3821 placebo tablets, Single administration
  Interventions: Drug: TQH3821 tablets (Placebo)
- TQH3821 Tablets (Food Effect) (Experimental): TQH3821 tablets, 2 sequential periods (fasting and fed)
  Interventions: Drug: TQH3821 tablets
- TQH3821 Placebo Tablets (Food Effect) (Placebo Comparator): TQH3821 placebo tablets, 2 sequential periods (fasting and fed)
  Interventions: Drug: TQH3821 tablets (Placebo)
- TQH3821 Tablets (Multiple Administration Dose) (Experimental): TQH3821 tablets once every 12 hours for 7 times during the continuous administration phase.
  Interventions: Drug: TQH3821 tablets
- TQH3821 Placebo Tablets (Multiple Administration Dose) (Placebo Comparator): TQH3821 placebo tablets once every 12 hours for 7 times during the continuous administration phase.
  Interventions: Drug: TQH3821 tablets (Placebo)
- TQH3821 Tablets + Methotrexate Tablets (Experimental): Take Methotrexate Tablets once in the first cycle, take TQH3821 Tablets once every 12 hours in the second cycle for 6 times, and then TQH3821 Tablets + Methotrexate Tablets once in the third cycle.
  Interventions: Drug: TQH3821 tablets; Drug: Methotrexate tablets
- TQH3821 Placebo Tablets + Methotrexate Tablets (Placebo Comparator): Take Methotrexate Tablets once in the first cycle, take TQH3821 placebo tablets once every 12 hours in the second cycle for 6 times, and then TQH3821 placebo tablets + Methotrexate Tablets once in the third cycle.
  Interventions: Drug: TQH3821 tablets (Placebo); Drug: Methotrexate tablets

INTERVENTIONS:
Drug: TQH3821 tablets — TQH3821 tablets is an Interleukin-1 receptor-associated kinase 4 inhibitor that exhibits a high degree of inhibitory activity against IRAK4 kinase.
  Arms: TQH3821 Tablets (Food Effect); TQH3821 Tablets (Multiple Administration Dose); TQH3821 Tablets (Single Administration Dose); TQH3821 Tablets + Methotrexate Tablets
Drug: TQH3821 tablets (Placebo) — TQH3821 tablets (Placebo) is a placebo produced with reference to TQH3821 tablets, which has no effect on IRAK4 kinase.
  Arms: TQH3821 Placebo Tablets (Food Effect); TQH3821 Placebo Tablets (Multiple Administration Dose); TQH3821 Placebo Tablets (Single Administration Dose); TQH3821 Placebo Tablets + Methotrexate Tablets
Drug: Methotrexate tablets — Methotrexate tablets is a folic acid antagonist, which belongs to an anti-rheumatic drug to improve the condition
  Arms: TQH3821 Placebo Tablets + Methotrexate Tablets; TQH3821 Tablets + Methotrexate Tablets

SUMMARY:
This study was a randomized, double-blind, placebo-controlled phase I clinical trial of TQH3821 in adult healthy subjects, which plans to recruit 72 healthy subjects.

The main purpose was to evaluate the safety and tolerance of different doses of TQH3821 or in combination with methotrexate tablets after single and multiple administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1 Sign an informed consent form before the test, and fully understand the content, process and possible adverse reactions of the test;
* 2 Be able to complete the research according to the requirements of the plan;
* 3 Subjects (including partners) are willing to voluntarily take effective contraception within 6 months from screening to the last study drug administration;
* 4 Male and female subjects aged 18 to 55 years (including critical value);
* 5 Male subjects weigh not less than 50 kg, female subjects weigh not less than 45 kg, BMI in the range of 18 ~ 28 kg / m2 (including critical value);
* 6 Physical examination, normal or abnormal vital signs are of no clinical significance

Exclusion Criteria:

* 1 Those who smoke more than 5 cigarettes per day in the 12 weeks before screening;
* 2 Allergic constitution (a variety of drug and food allergies);
* 3 Have a history of substance abuse, drug and/or alcohol abuse;
* 4 Donate blood or lose a lot of blood (> 450 mL) within 12 weeks prior to screening;
* 5 Take any drug that alters the activity of liver enzymes 28 days before screening, or combined with inhibitors or inducers of Cytochrome P4503A4 enzyme (CYP3A4 );
* 6 Took any prescription drugs, over-the-counter drugs, any vitamin products or herbs within 14 days prior to screening;
* 7 Those who have taken a special diet or have strenuous exercise within 2 weeks before screening, or other factors that affect drug absorption, distribution, metabolism, excretion and other factors;
* 8 Those who are vaccinated with live attenuated vaccines within 28 days before the start of research treatment, inactivated vaccines within 7 days, or vaccinated during the study period;
* 9 Have taken research drugs within 12 weeks before taking our research drugs, or participated in clinical trials of drugs;
* 10 Have a history of dysphagia or any gastrointestinal diseases that affect the absorption of the drug or a history of gallbladder resection or biliary tract diseases;
* 11 Have any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or stomach and duodenal ulcers;
* 12 Subjects who could not tolerate a standard meal; (only applies to subjects participating in the postprandial test);
* 13 Electrocardiogram (ECG) abnormalities have clinical significance;
* 14 Female subjects are breastfeeding during the screening period or during the test or have a positive serum pregnancy result;
* 15 Diseases with abnormal clinical significance in clinical laboratory examination or other clinical findings within 24 weeks before screening;
* 16 Positive screening for viral hepatitis (including hepatitis B and C), Acquired Immune Deficiency Syndrome (AIDS) antibodies, treponemal antibodies;
* 17 Acute illness or concomitant medication from the screening stage to the study of medication;
* 18 Chocolate, any caffeinated or xanthine-rich foods or beverages taken 24 hours before taking the study drug;
* 19 Have taken any products containing alcohol within 24 hours before taking the research medication;
* 20 Positive for urine drug screening;
* 21 Participants who were considered by the investigators to have other factors that were not suitable for this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | The first day of the first administration until 8 days after the last administration
  Safety and tolerability are assessed by the incidence of adverse events and its severity caused by the study drug during or after dose.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Pharmacokinetics blood samples were collected from 60 minutes before administration on Day 1 to 168 hours after the last administration.
  Peak concentration (Cmax) refers to the highest blood drug concentration achieved after administration called blood drug peak concentration (referred to as peak concentration), which is related to the dose administered, the route of administration, the number of times of administration and the time of arrival
Plasma concentration-area under time curve (AUC0-t) | Pharmacokinetics blood samples were collected from 60 minutes before administration on Day 1 to 168 hours after the last administration.
  The area under the plasma concentration-time curve from the beginning of the first administration to the last measurable concentration point
Plasma concentration-area under time curve (AUC0-∞) | Pharmacokinetics blood samples were collected from 60 minutes before administration on Day 1 to 168 hours after the last administration.
  Extrapolated from the first administration to the area under the plasma concentration-time curve to infinity
High sensitivity C-reactive protein (hs-CRP) | Multiple Administration Dose: Blood samples were collected from 60 minutes before administration on Day 1 to 192 hours after the consecutive administration.
  Hypersensitive C-reactive protein is a kind of C-reactive protein in plasma. It is a non-specific marker of acute systemic inflammatory response synthesized by the liver

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China